CLINICAL TRIAL: NCT07065890
Title: Association Between Body Roundness Index and Wound Healing Post-Thoracic Surgery: A Prospective Study
Brief Title: Association Between Body Roundness Index and Wound Healing
Status: Completed | Type: Observational
Sponsor: Zhao bo (Other)
Responsible Party: Sponsor-Investigator, Zhao bo, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-JRB202503009
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Thoracic Surgery; Obesity; BMI; Visceral Fat; Wound Healing
Keywords: BRI; Thoracic Surgery; Wound Healing; BMI; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- impaired wound healing: This cohort include individuals diagnosed with poor wound healing according to the definitions and guidelines for assessment of wounds and evaluation of healing

SUMMARY:
Background Obesity is a significant risk factor for adverse postoperative outcomes, including impaired wound healing. This study aimed to investigate the association between the Body Roundness Index (BRI) and impaired wound healing following thoracic surgery.

Methods This study included 387 patients who underwent thoracic surgery at Tongji Hospital in Wuhan between October 2024 and January 2025. Wound healing was assessed 30 days postoperatively. Logistic regression and propensity score matching (PSM) analyses were performed to evaluate the relationship between BRI and impaired wound healing, with subgroup analyses conducted to further explore this association.

DETAILED DESCRIPTION:
This prospective cohort study collected clinical data from patients undergoing thoracic surgery at Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, between October 1, 2024, and January 30, 2025. Initial enrollment included 422 patients, with 387 participants retained after data cleaning (Figure 1). The primary objective was to evaluate the association between BRI and impaired postoperative wound healing through multivariable logistic regression, propensity score matching (PSM), and subgroup analyses.

ELIGIBILITY:
Inclusion Criteria：

* Patients who underwent surgical treatment in the Department of Thoracic Surgery at Tongji Hospital;
* Complete clinical data and diagnostic test results available;
* Postoperative follow-up conducted regularly in accordance with medical advice, with comprehensive follow-up records；

Exclusion Criteria:

* Without surgery or transferred to other departments；
* Missing basic information；
* Failure to review on time or refusal to follow up；
* Additional surgeries within 30 days of discharge from the hospital；

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study collected clinical data from patients undergoing thoracic surgery at Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, between October 1, 2024, and January 30, 2025. Initial enrollment included 422 patients, with 387 participants retained after data cleaning.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Wound healing | From the day of surgery to 30 days postoperatively
  Determine the presence of impaired wound healing based on the definitions and guidelines for wound assessment and evaluation of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang q Zhang, Dr., Study Director — Tongji Medical College of HUST Tongji Medical College Tongji Hospital
Locations (1):
- Tongji Medical College of HUST Tongji Medical College Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT07065890/Prot_000.pdf